CLINICAL TRIAL: NCT05074732
Title: Dundrum Forensic Redevelopment Evaluation Study: D-FOREST Study.
Acronym: D-FOREST
Status: Recruiting | Type: Observational
Sponsor: Health Service Executive, Ireland (Other)
Responsible Party: Principal Investigator, Dr Mary Davoren, Consultant Forensic Psychiatrist and Clinical Senior Lecturer in Forensic Psychiatry, Health Service Executive, Ireland
Other Study IDs: HSEIreland
Record Dates: First submitted 2021-10-02; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Schizophrenia; Forensic Psychiatry; Outcome Measure; Violence; Personality Disorders; Recovery; Obesity; Type II Diabetes; Cardiovascular Diseases; Frailty; Psychosis; Treatment-resistant Schizophrenia
MeSH Terms: conditions — Schizophrenia; Personality Disorders; Obesity; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Frailty; Psychotic Disorders; Schizophrenia, Treatment-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The DUNDRUM Forensic Redevelopment Evaluation study (D-FOREST study) is a multi-site comprehensive evaluation of a complete National Forensic Mental Health Service. The study will have a prospective, observational, longitudinal design which will permit the evaluation of benefit over time for individual patients, groups of patients and the evaluation of the benefit in terms of service based outcomes of the redevelopment of a complete National Forensic Mental Health Service e.g. effects on waiting list times, length of stay. The study will systematically evaluate multiple domains of recovery in a complete National Forensic Service, including patients' physical health, mental health, offending behaviours and social and occupational functioning.

DETAILED DESCRIPTION:
The DUNDRUM Forensic Redevelopment Evaluation Study (D-FOREST).

Forensic Mental Health Services have a dual role, to treat mental disorder and reduce violent recidivism. Forensic mental health services are low volume, high cost services and therefore it is vital to conduct robust outcome measure studies to demonstrate benefit and effectiveness. D-FOREST is a study comprising the evaluation of a complete national forensic mental health service at a time of significant change, that of the re-development of Ireland's National Forensic Mental Health Service from a 19th century building to a complete national service in North Dublin.

We hypothesise that the redevelopment of the campus from Dundrum Hospital to a new 170-bed hospital in Portrane will demonstrate improvements in two main areas, firstly service wide improvements and secondly patient benefit related improvements.

We hypothesise that the development of the new campus at Portrane will lead to reduced time on the waiting list for admission and reduced length of stay in the hospital as well as sustainable rates of admissions and discharges maintained over the five year period of this study.

We anticipate that the newly expanded hospital will be able to facilitate the admission of patients with higher security needs from the prison settings, and therefore there may be a rise in the security needs profile of the group, while urgency of need for admission on the waiting list will decrease.

We anticipate that patient engagement with group and individual therapy will improve with greater access to therapists as the staff number will expand and therefore measures of therapeutic programme completion and recovery and measures of risk in a broad sense should improve across the patient group. We also anticipate finding improved measures of patient ratings on environmental measures such as ward atmosphere on moving to the new campus.

Repeated measures in the area of physical health, mental health and violence risk and forensic recovery will be taken, at baseline (time of admission to the service) as well as at six-monthly intervals throughout the patients admission journey. These main areas will include structured interview measures of psychopathology e.g. SCID, PANSS, clinician rated measures violence and self-harm risk assessment instruments e.g. HCR-20, SRAMM, and measures of therapeutic programme completion and recovery (DUNDRUM-3 and DUNDRUM-4 scales) as well as overall functioning MIRECC GAF. Physical health measures will include measures of BMI, frailty and sedentary behaviours.

Other measures including ward atmosphere scales ESSENCES and measures of quality of life (WHO-QUOL) will also be offered to the patient group to complete.

A combination of both self-rated and interview based measures to engage patients, and clinician rated measures will be used. This is due to the high rates of treatment resistant psychoses in forensic hospital settings, and therefore to rely on self-rated or interview rated measures along would mean that many of the most unwell patients may not be able or willing to engage. Thus utilising this combination approach ensures that any bias in the results and outcomes observed will be minimised.

Statistical analysis plan:

Statistical methods for primary and secondary outcomes. Time intervals (time in days to admission from waiting list, length of stay) will be measured by median and 95% confidence interval using Kaplan Meyer and Cox regression analyses. Survival analysis will be used to assess factors affecting length of stay.

Patient level measures will be expressed as changes from baseline (typically from the time of admission) using ANCOVA, MANOVA or logistic regression as appropriate with correction for the effects of static baseline variables such as demographic characteristics (e.g. age, sex and ethnicity) or diagnosis including multi-axial diagnoses, neurocognitive function, and legal status. Measures of effect size will be used alongside measures of statistical significance for primary and secondary outcomes. At the individual level measures of reliable and clinically meaningful change will be calculated and proportions achieving this will be expressed with 95% confidence intervals.

Analysis of repeated measures will be used to compare mean scores on measures of physical health, risk of violence, therapeutic programme completion, recovery and overall functioning, at time points in advance of the move of the NFMHS to the new Portrane Hospital Campus and for five years after the move.

Lagged causal model analysis will be used to assess the existence and significance of potential directed relationships between the baseline measures of symptomatology of schizophrenia and violence risk and final outcome namely length of stay.

The lagged causal model approach will be used also to examine the relationship between amount of 'treatment' received and change in outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the National Forensic Mental Health Service (NFMHS) Ireland after 1st December 2019 until 7 years after the transfer of the National Service to the newly developed complete National Forensic Service at Portrane, North Dublin, Ireland.

Exclusion Criteria:

* This study comprises a complete cohort of admissions to the NFMHS. All adult patients admitted during the time period will be included in the study, regardless of their length of stay.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The NFMHS Ireland provides secure forensic mental health services for adult men and women, who require care and treatment in conditions of therapeutic security.
  All patients are over 18 years. The majority of patients will have a major mental illness, most commonly treatment resistant schizophrenia, with high rates of polysubstance misuse, personality co-morbidity and physical health issues such as obesity and type II diabetes.
  All patients are deemed to pose a serious risk of violence towards others. All patients are detained under mental health legislation, with over 40% having been found not guilty by reason of insanity (not criminally responsible due to illness) of a serious offence.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Length of stay in the secure forensic hospital setting. | 5 years
  Length of stay in the secure forensic hospital setting
Recovery from psychosis | 5 years
  Reduction in psychotic symptoms and stabilisation of psychosis
Reduction in violence | 5 years
  Reduction in violent behaviours, violent incidents and pro-violent attitudes

SECONDARY OUTCOMES:
Reducing BMI and sedentary behaviours | 5 years
  Improving physical health measures namely reduction in obesity and reduction in sedentary behaviours
Improving overall functioning level | 5 years
  Improving scores on GAF MIRECC for measure of overall functioning

CONTACTS AND LOCATIONS:
Overall Officials: Mary Davoren, M.D., Principal Investigator — Trinity College University of Dublin
Locations (1):
- National Forensic Mental Health Service, Central Mental Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
Due to the uniquely sensitive nature of data from secure forensic mental health services, aggregate anonymised data only will be presented and published. Any access to aggregated anonymised datasets will be considered by request on a case-by-case basis only.

REFERENCES:
- [Background] Davoren M, Abidin Z, Naughton L, Gibbons O, Nulty A, Wright B, Kennedy HG. Prospective study of factors influencing conditional discharge from a forensic hospital: the DUNDRUM-3 programme completion and DUNDRUM-4 recovery structured professional judgement instruments and risk. BMC Psychiatry. 2013 Jul 9;13:185. doi: 10.1186/1471-244X-13-185. PMID 23837697
- [Background] Davoren M, O'Dwyer S, Abidin Z, Naughton L, Gibbons O, Doyle E, McDonnell K, Monks S, Kennedy HG. Prospective in-patient cohort study of moves between levels of therapeutic security: the DUNDRUM-1 triage security, DUNDRUM-3 programme completion and DUNDRUM-4 recovery scales and the HCR-20. BMC Psychiatry. 2012 Jul 13;12:80. doi: 10.1186/1471-244X-12-80. PMID 22794187
- [Background] Donnelly V, Lynch A, Devlin C, Naughten L, Gibbons O, Mohan D, Kennedy HG. Therapeutic alliance in forensic mental health: coercion, consent and recovery. Ir J Psychol Med. 2011 Mar;28(1):21-28. doi: 10.1017/S0790966700011861. PMID 30199989
- [Background] Davoren M, Fitzpatrick M, Caddow F, Caddow M, O'Neill C, O'Neill H, Kennedy HG. Older men and older women remand prisoners: mental illness, physical illness, offending patterns and needs. Int Psychogeriatr. 2015 May;27(5):747-55. doi: 10.1017/S1041610214002348. Epub 2014 Nov 27. PMID 25428523
- [Background] Donnelly V, Lynch A, Mohan D, Kennedy HG. Working alliance, interpersonal trust and perceived coercion in mental health review hearings. Int J Ment Health Syst. 2011 Nov 10;5(1):29. doi: 10.1186/1752-4458-5-29. PMID 22074788
- [Background] Ijaz A, Papaconstantinou A, O'Neill H, Kennedy HG. The Suicide Risk Assessment and Management Manual (S-RAMM) Validation Study 1. Ir J Psychol Med. 2009 Jun;26(2):54-58. doi: 10.1017/S0790966700000215. PMID 30282262
- [Background] Flynn G, O'Neill C, McInerney C, Kennedy HG. The DUNDRUM-1 structured professional judgment for triage to appropriate levels of therapeutic security: retrospective-cohort validation study. BMC Psychiatry. 2011 Mar 16;11:43. doi: 10.1186/1471-244X-11-43. PMID 21410967
- [Background] Freestone M, Bull D, Brown R, Boast N, Blazey F, Gilluley P. Triage, decision-making and follow-up of patients referred to a UK forensic service: validation of the DUNDRUM toolkit. BMC Psychiatry. 2015 Oct 7;15:239. doi: 10.1186/s12888-015-0620-9. PMID 26446536
- [Background] Kennedy H, O'Neill C, Flynn G, Gill P, Davoren M. The DUNDRUM toolkit draft V1. 0.30. Dublin: Trinity College Dublin; 2016.
- [Background] Kennedy, H. (2021). Models of care in forensic psychiatry. BJPsych Advances, 1-14. doi:10.1192/bja.2021.34
- [Result] Williams HK, Senanayke M, Ross CC, Bates R, Davoren M. Security needs among patients referred for high secure care in Broadmoor Hospital England. BJPsych Open. 2020 Jun 2;6(4):e55. doi: 10.1192/bjo.2020.35. PMID 32482202
- [Result] Kennedy HG, Mullaney R, McKenna P, Thompson J, Timmons D, Gill P, O'Sullivan OP, Braham P, Duffy D, Kearns A, Linehan S, Mohan D, Monks S, McLoughlin L, O'Connell P, O'Neill C, Wright B, O'Reilly K, Davoren M. A tool to evaluate proportionality and necessity in the use of restrictive practices in forensic mental health settings: the DRILL tool (Dundrum restriction, intrusion and liberty ladders). BMC Psychiatry. 2020 Oct 23;20(1):515. doi: 10.1186/s12888-020-02912-6. PMID 33097036
- [Result] Basrak N, Mulcrone N, Sharifuddin S, Ghumman Z, Bechan N, Mohamed E, Murray M, Rajendran H, Gunnigle S, Nolan M, Quane T, Terao M, Hoare T, Kirrane K, Kennedy HG, Davoren M. Risk of adverse outcome of COVID-19 among patients in secure psychiatric services: observational cohort study. BJPsych Open. 2021 Jan 11;7(1):e31. doi: 10.1192/bjo.2020.169. PMID 33427191
- [Result] Davoren M, Byrne O, O'Connell P, O'Neill H, O'Reilly K, Kennedy HG. Factors affecting length of stay in forensic hospital setting: need for therapeutic security and course of admission. BMC Psychiatry. 2015 Nov 23;15:301. doi: 10.1186/s12888-015-0686-4. PMID 26597630
- [Result] Abidin Z, Davoren M, Naughton L, Gibbons O, Nulty A, Kennedy HG. Susceptibility (risk and protective) factors for in-patient violence and self-harm: prospective study of structured professional judgement instruments START and SAPROF, DUNDRUM-3 and DUNDRUM-4 in forensic mental health services. BMC Psychiatry. 2013 Jul 27;13:197. doi: 10.1186/1471-244X-13-197. PMID 23890106
- [Derived] Davoren M, O'Reilly K, Mohan D, Kennedy HG. Prospective cohort study of the evaluation of patient benefit from the redevelopment of a complete national forensic mental health service: the Dundrum Forensic Redevelopment Evaluation Study (D-FOREST) protocol. BMJ Open. 2022 Jul 22;12(7):e058581. doi: 10.1136/bmjopen-2021-058581. PMID 35868830